CLINICAL TRIAL: NCT06848816
Title: DUTRAPYL STUDY : Duration of Antibiotic Therapy in Acute Kidney Graft Pyelonephritis: Effect on the Risk of Recurrence
Brief Title: Duration of Antibiotic Therapy in Acute Kidney Graft Pyelonephritis (AGPN): Effect on the Risk of Recurrence
Acronym: DUTRAPYL
Status: Active, not recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, CORBEL Alice, M.D., Central Hospital, Nancy, France
Other Study IDs: DUTRAPYL
Record Dates: First submitted 2025-02-16; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pyelonephritis Acute; Kidney Transplantation Recipients
Keywords: Acute graft pyelonephritis; duration treatment; antibiotic; recurrence; relapse
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to evaluate the impact of the duration of antibiotic therapy on the risk of recurrence in kidney graft pyelonephritis. The secondary objectives are to identify the factors associated with the duration of antibiotic therapy in acute kidney graft pyelonephritis, identify the factors associated with recurrence of acute kidney graft pyelonephritis within 3 months, evaluate the impact of the duration of antibiotic therapy on antibiotic-related complications and assess the impact of the duration of antibiotic therapy on the progression of renal function after acute kidney graft pyelonephritis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Kidney transplant recipients with a functional graft.
* Hospitalization with acute pyelonephritis (APN) defined by fever OR chills (noted in the clinical records) AND bacteriuria AND exclusion of another obvious cause of fever. (For rehospitalizations, also include cases where antibiotic therapy was initiated based on suspicion, even in the absence of documented infection.)

Exclusion Criteria:

* Age < 18 years.
* Vacationing patient or lost to follow-up with follow-up < 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient with AGPN during the study period
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relaspe AGPN | 3 month
  Rehospitalization for acute kidney graft pyelonephritis (AGPN) within three months after completion of treatment

SECONDARY OUTCOMES:
Early AGPN relapse | 1 month
  Rehospitalization for acute kidney graft pyelonephritis (AGPN) within one month after completion of treatment
ITU relapse | 3 month
  Antibiotic treatment for urinary tract infection within 3 months after completion of treatment.
Identical microorganism relapsing AGPN | 3 month
  New episode of AGPN with the same pathogen within 3 months after completion of treatment
Multidrug resistant emerging pathogens | 3 month
  Infection with a multidrug-resistant bacteria within 3 months after completion of treatment
Clostridioides difficile colitis | 3 month
  Occurrence of Clostridioides difficile colitis within 3 months after completion of treatment
Early kidney function evolution | 1 month
  Evolution of renal function (creatininemia) 1 month after completion of treatment for APNAG.
3 month kidney function evolution | 3 month and 21 days
  Evolution of renal function (creatininemia) 3 +/- 21 days after completion of treatment for AGPN
Risk factors | 3 month
  Clinical and biological Factors associated with AGPN recurrence independently of the duration of antibiotic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided